CLINICAL TRIAL: NCT00116363
Title: Phase II Study Examining the Biological Efficacy of Intratumoral INGN 241 (Ad-mda7) Administration in Patients With In Transit Melanoma
Brief Title: Safety and Efficacy Study of INGN 241 Gene Therapy in Patients With In Transit Melanoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Introgen Therapeutics (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 241-004; 2003-0590, R43 CA 89778
Expanded Access: Available
Record Dates: First submitted 2005-06-28; First posted 2005-06-29 (Estimated); Last update posted 2008-04-01 (Estimated); Status verified 2008-03

CONDITIONS: Malignant Melanoma; Neoplasm Metastasis
Keywords: gene therapy; melanoma; adenovirus; in-transit melanoma; metastatic melanoma
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Adenoviridae Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: investigational drug INGN 241

SUMMARY:
This is a research study to look at the ways in which a treatment called INGN241 can kill melanoma cells or help the patient's immune system kill melanoma cells.

DETAILED DESCRIPTION:
INGN 241 is an adenoviral vector carrying the MDA-7 cDNA. MDA-7 is a novel tumor suppressor molecule with cytokine properties, recently designated as IL-24. Over expression of MDA-7 in melanoma cells in vitro has been shown to inhibit cellular proliferation and induce apoptosis. Loss of MDA-7 expression in human melanomas has been shown to correlate with invasion and metastasis. The INGN 241 gene transfer construct has been previously used in human subjects in an ongoing open label Phase I study using intratumoral administration, and has been well tolerated to date. The primary objectives of the present study are to determine if INGN 241, injected into a melanoma in transit lesion, can induce apoptosis in regional uninjected lesions and initiate systemic immune activation. Secondary objectives include examination of specific immunity and of clinical response and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven melanoma, must have 3 regional metastatic lesions that are in transit

Exclusion Criteria:

* Central nervous system involvement by melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2005-03; Study Completion 2006-12 (Estimated)

PRIMARY OUTCOMES:
anti-tumor effects and systemic immune activation at 28 days

SECONDARY OUTCOMES:
tumor response
toxicity and safety
the induction of antigen-specific T-lymphocytes after multiple cycles of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin B Kim, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Casciello F, Kelly GM, Ramarao-Milne P, Kamal N, Stewart TA, Mukhopadhyay P, Kazakoff SH, Miranda M, Kim D, Davis FM, Hayward NK, Vertino PM, Waddell N, Gannon F, Lee JS. Combined Inhibition of G9a and EZH2 Suppresses Tumor Growth via Synergistic Induction of IL24-Mediated Apoptosis. Cancer Res. 2022 Apr 1;82(7):1208-1221. doi: 10.1158/0008-5472.CAN-21-2218. PMID 35149587